CLINICAL TRIAL: NCT05122130
Title: Effect of Topically Applied Melatonin (N-ACETYL-5-METHOXY TRYPTAMINE) Loaded Gelatin Sponge on Palatal Wound Healing (Randomized Controlled Clinical Trial)
Brief Title: Effect of Melatonin on Palatal Wound Healing (Randomized Controlled Clinical Trial)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salma Nabil (Other)
Responsible Party: Sponsor-Investigator, Salma Nabil, principle investigator, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0252-06/2021
Record Dates: First submitted 2021-11-05; First posted 2021-11-16 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Wound Heal
Keywords: Gelatin sponge; melatonin
MeSH Terms: interventions — Melatonin; carboxypolymethylene

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study will be double-blinded where the patients and the statistician will be unaware of the treatment assignment till the end of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin group (Experimental): Melatonin loaded Carbopol hydrogel will be synthesized as follows: 1 gm of Carbopol will be dissolved in 100 ml deionized water while stirring at 600 rpm for 25°C. Melatonin (3gm) will be dissolved in 1 ml ethanol and added to the formed gel while stirring at 600 rpm at 25 °C. The pH will be adjusted to 7.4 using triethanolamine until a gel is formed and it will be loaded on gelatin sponge and will be applied to the donor site.
  Interventions: Drug: Melatonin
- Placebo group (Placebo Comparator): •Topical placebo carbopol gel will be prepared as follows: 1 gm of Carbopol will be dissolved in 100ml deionized water while stirring at 600 rpm for 25°C. The pH will be adjusted to 7.4 using triethanolamine until a gel is formed
  Interventions: Drug: Carbopol

INTERVENTIONS:
Drug: Melatonin — The donor site will be dressed with melatonin loaded gelatin sponge
  Other Names: N-ACETYL-5-METHOXY TRYPTAMINE
  Arms: Melatonin group
Drug: Carbopol — The donor site will be dressed with carbopol loaded gelatin sponge (placebo).
  Arms: Placebo group

SUMMARY:
The aim of the study is to assess the effect of topical melatonin loaded gelatin sponge on donor palatal site healing, after palatal graft harvesting.

DETAILED DESCRIPTION:
Autogenous soft tissue grafts can be considered the gold standard treatment for many muco-gingival problems. The most common site for harvesting soft tissue grafts is the palate. Many harvesting techniques have emerged, but the epithelialized graft harvesting technique is one of the most reliable and effective techniques as it imparts the superficial section of the connective tissue which contains the highest amount of lamina propria. Unfortunately, it leaves an open palatal wound healed by secondary intention, increasing pain and post-operative morbidity. In order to overcome these inadequacies investigators will cover the donor site with melatonin loaded gelatin sponge and evaluate its effect on the healing process.

ELIGIBILITY:
Inclusion Criteria

1. Patients who have at least one site of natural dentition or dental implants that need to be treated by free palatal graft surgery for indications including progressive recession, planned prosthodontics, presence of a mucogingival deformity, or a lack of keratinized gingiva.
2. Patients who have at least 4 mm thickness of palatal mucosa (at donor site)

Exclusion Criteria:

1. History of smoking.
2. Patients who have any known disease that interfere with periodontal surgery.
3. Patients who have any dermal or autoimmune diseases.
4. Patients who have any previous adverse reactions to the products (or similar products) used in this study.
5. Pregnant and lactating women.
6. Patients who have a palatal infection.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
palatal wound healing | Up to 2 weeks
  Standardized clinical photographs of the palatal surgical sites will be taken and will be imported into a software program (ImageJ 1.49v) and wound areas will be calculated by computerized planimetry (Difference in remaining wound area [mm2])

SECONDARY OUTCOMES:
Intensity of pain | Up 2 weeks
  by visual analogue scale Patients will be asked to grade the severity of their symptoms on VAS that ranges from (0-100 mm)

CONTACTS AND LOCATIONS:
Overall Officials: salma Nabil, BDS, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt